CLINICAL TRIAL: NCT00490087
Title: Operational Hysteroscopy Versus Traditional Surgery: Costs and Health Benefits
Brief Title: Resectoscopic Treatment of Atypical Endometrial Polyps in Fertile Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC 23/98
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2007-06

CONDITIONS: Atypical Endometrial Polyps; Atypical Endometrial Hyperplasia
Keywords: Atypical endometrial polyps; Atypical Endometrial Hyperplasia; Hysteroscopic resection; Conservative treatment; Fertile women
MeSH Terms: conditions — Endometrial Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hysteroscopic resection plus IUD (Experimental)
  Interventions: Device: Levonorgestrel intrauterine device (IUD)
- Hysteroscopic resection without IUD (No Intervention)

INTERVENTIONS:
Device: Levonorgestrel intrauterine device (IUD)
  Arms: Hysteroscopic resection plus IUD

SUMMARY:
The study aims to evaluate the long-term efficacy and prognosis of hysteroscopic resection and coagulation of the base of endometrial polyps with focal atypia in fertile women.

DETAILED DESCRIPTION:
The introduction of hysteroscopy in clinical practice changed significantly our knowledge of uterine cavity, but did not stimulate the start of big studies with aim to evaluate the feasibility of conservative treatments for better defined diseases as endometrial polyp. The use of curettage(D&C) has led the gynecologists to consider diffuse atypical endometrial hyperplasia and atypical polyp as the same disease. The treatment of these precancerous lesions recommended by scientific societies is aggressive (hysterectomy). Surprisingly, regarding hysterectomy we did not observe management modifications after the introduction of endoscopic techniques, as happened in other surgical disciplines.

To evaluate costs and health benefits of operational hysteroscopy we started in our Institute a study protocol in 1998. In a first trial we studied a conservative treatment of postmenopausal woman with high anesthesiologic risk who had endometrial polyps with atypia and no involvement of the base (Scrimin F. Am J Obstet Gynecol 2006;195:1328-30).

The good initial results and the request of conservative treatments by some women, desiring pregnancies, encouraged us to start this preliminary trial to evaluate the long-term efficacy and prognosis of hysteroscopic resection and coagulation of the base of endometrial polyps with focal atypia in a little sample of fertile women. Other studies suggest progestin treatment of well differentiated carcinoma in young women who desired to preserve their fertility. There is no evidence of a correlation between the tendency to develop endometrial polyps and the risk of endometrial carcinoma. The risk of malignant degeneration of endometrial polyps is not well known, but seems to range between 0.5% and 6%. On this background, we decided to study in the same population of fertile women and with a quasi-randomised design the possible additional effect of levonorgestrel-releasing intrauterine device (LNG-IUD).

Comparison: women assigned to odd numbers underwent polyp resection and endometrial surveillance with insertion of levonorgestrel intrauterine system (IUD group), women assigned to even numbers underwent polyp resection and endometrial surveillance without insertion of levonorgestrel intrauterine system (no IUD or control group).

ELIGIBILITY:
Inclusion Criteria:

* women in fertile age desiring to preserve their uterus
* atypical polyps, without atypia in the base. The hysteroscopic and histologic criteria for inclusion in the study were: proliferative, secretive, dysfunctional endometrium or simple hyperplasia in 4 random biopsies.

Exclusion Criteria:

* women with adenomatous or atypical hyperplasia in the random biopsies

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 1999-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Efficacy and prognosis of hysteroscopic resection of atypical polyps in terms of appearance of endometrial cancer or recurrence of atypical endometrial lesions | Five years

SECONDARY OUTCOMES:
Recurrence rate of polyp in the two groups | Five years

CONTACTS AND LOCATIONS:
Overall Officials: Federica Scrimin, MD, Principal Investigator — Institute of Child Health IRCCS Burlo Garofolo, Trieste, Italy
Locations (1):
- Institute of Child Health, IRCCS Burlo Garofolo, Trieste, Friuli Venezia Giulia, Italy

REFERENCES:
- [Result] Scrimin F, Wiesenfeld U, Candiotto A, Inglese S, Ronfani L, Guaschino S. Resectoscopic treatment of atypical endometrial polyps in fertile women. Am J Obstet Gynecol. 2008 Oct;199(4):365.e1-3. doi: 10.1016/j.ajog.2008.03.041. PMID 18928975